CLINICAL TRIAL: NCT00377936
Title: A Controlled, Randomized, Open Label Phase II Trial to Evaluate Safety and Efficacy of a 1st Line Combination Treatment With Weekly Infusions of Gemcitabine and Twice Weekly Administration of Lipid Complexed Paclitaxel (EndoTAG-1) in Three Dose Levels Compared With Gemcitabine Monotherapy in Patients With Measurable Locally Advanced and/or Metastatic Adenocarcinoma of the Pancreas
Brief Title: EndoTAG-1 / Gemcitabine Combination Therapy to Treat Locally Advanced and/or Metastatic Adenocarcinoma of the Pancreas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MediGene (Industry)
Responsible Party: Susanne Kienzle-Horn / Clinical Trial Manager, MediGene
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT4001; EudraCT No.: 2005-000666-39
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Last update posted 2008-11-14 (Estimated); Status verified 2008-11

CONDITIONS: Adenocarcinoma; Metastasis; Pancreas Neoplasms
Keywords: Adenocarcinoma of the pancreas; Locally advanced; Metastatic
MeSH Terms: conditions — Adenocarcinoma; Neoplasm Metastasis; Pancreatic Neoplasms | interventions — Gemcitabine; MBT-0206

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Gemcitabine
  Interventions: Drug: Gemcitabine alone
- 2 (Experimental): EndoTag-1 + Gemcitabine
  Interventions: Drug: EndoTAG-1 and Gemcitabine
- 3 (Experimental): EndoTag-1 + Gemcitabine
  Interventions: Drug: EndoTAG-1 and Gemcitabine
- 4 (Experimental): EndoTag-1 + Gemcitabine
  Interventions: Drug: EndoTAG-1 and Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine alone — Gemcitabine monotherapy 1000 mg/m2 weekly
  Arms: 1
Drug: EndoTAG-1 and Gemcitabine — EndoTAG-1 11 mg/m2 twice weekly + Gemcitabine 1000 mg/m2 weekly
  Arms: 2
Drug: EndoTAG-1 and Gemcitabine — EndoTAG-1 22 mg/m2 twice weekly + Gemcitabine 1000 mg/m2 weekly
  Arms: 3
Drug: EndoTAG-1 and Gemcitabine — EndoTAG-1 44 mg/m2 twice weekly + Gemcitabine 1000 mg/m2 weekly
  Arms: 4

SUMMARY:
The intention of this trial is to evaluate safety and efficacy of a combination treatment of EndoTAG-1 with Gemcitabine versus Gemcitabine monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Inoperable adenocarcinoma of the pancreas
* Histologic or cytologic confirmation
* At least 18 years of age

Exclusion Criteria:

* Any chemotherapeutical treatment for pancreatic adenocarcinoma before enrollment
* Major surgery within 4 weeks prior to enrollment
* Major cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2005-09; Primary Completion 2008-06 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival | Median
6-month-survival-rate | 6 Months
Overall survival | Median

SECONDARY OUTCOMES:
Incidence and percentage of patients with Adverse Events | 28 days after last patient out
Number of clinically significant abnormal laboratory values | Last patient out

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Löhr, Prof., Principal Investigator — Universitätsklinikum Mannheim
Locations (3):
- Prague, Czechia
- Budapest, Hungary
- Kiev, Ukraine